CLINICAL TRIAL: NCT07301892
Title: Impact of Generative Artificial Intelligence on Diagnosing Rheumatoid Arthritis Complications
Brief Title: Generative AI Impact on Rheumatoid Arthritis Complications Diagnosis
Status: Recruiting | Type: Observational
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Quan Jiang, Director of the Rheumatology Department, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Other Study IDs: 2025-201-KY
Record Dates: First submitted 2025-09-28; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Rheumatoid Arthritis (RA; Osteoporosis; Osteoarthritis; Interstitial Lung Disease; Thyroid Diseases; Cardiovascular Diseases; Pulmonary Complications; Sjogren's Syndrome; Liver Disorders; Renal Lesions; Vasculitis; Amyloidosis; Peripheral Neuropathy; Thrombosis; RA Complications
Keywords: Rheumatoid Arthritis; generative AI; large language model; Rheumatoid arthritis complications
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoporosis; Osteoarthritis; Lung Diseases, Interstitial; Thyroid Diseases; Cardiovascular Diseases; Sjogren's Syndrome; Digestive System Diseases; Vasculitis; Amyloidosis; Peripheral Nervous System Diseases; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RA patient group using generative AI prediction reports: Inpatients newly diagnosed with rheumatoid arthritis in our rheumatology department between October 1, 2025, and June 2026 will be recruited for the study. Physicians will use GenAI predictions of potential RA complications and co-existing diseases, together with confirmatory diagnostic tests, as additional inputs in the differential diagnosis process.
  Interventions: Other: Generative AI prediction report for RA complications

INTERVENTIONS:
Other: Generative AI prediction report for RA complications — Generative AI based on multiple large language models (LLMs) is used to predict potential complications and co-existing diseases in patients with rheumatoid arthritis using EHR data available at admission. Physicians use these AI predictions as additional information to adjust their diagnostic plans during differential diagnosis. The impact of this intervention on the final diagnoses at discharge will be measured.
  Before the prospective study, the adoptability of the generative AI prediction reports will be validated using EHR records from retrospective RA patients.

SUMMARY:
Generative AI (GenAI) based on large language models (LLMs) is expected to improve the diagnosis and treatment of autoimmune diseases. We are studying how GenAI may affect the diagnosis of various complications of rheumatoid arthritis (RA). In a retrospective study using RA patients' EHR records, we will quantify physician adoption of GenAI predictions for RA complications and co-existing diseases. In a prospective observational study, we will assess the feasibility of using GenAI predictions as additional clinical information to help physicians make more complete diagnoses of RA complications and co-existing diseases, including complex, uncommon, or rare conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an initial diagnosis of rheumatoid arthritis (RA).
* All real-world RA inpatients admitted to our department.
* Admission occurring within the real-world data study period.

Exclusion Criteria:

* Patients subsequently confirmed not to have RA during the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult male and female RA inpatients admitted to our Rheumatology Department who fulfill the 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) classification and diagnostic criteria for rheumatoid arthritis.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Will physicians adopt GenAI predictions in diagnosing RA complications? | Immediately after reviewing patient AI report on the day of admission.
  In the routine care workflow, large language models (LLMs) are used to predict potential RA complications for each de-identified patient case and generate an AI report listing possible complications and co-existing diseases. Additional diagnostic tests are suggested to verify the predicted conditions. After reviewing the AI report, physicians immediately evaluate each disease prediction using a 5-point Likert scale (1 = complete disagreement; 2 = disagreement; 3 = neutral; 4 = agreement; 5 = complete agreement). The mean score is calculated as a measure of perceived prediction accuracy. Physicians also indicate whether each specific disease prediction could potentially be adopted or used to assist differential diagnosis (binary: 0 or 1). The percentage of positive adoption responses is calculated as a measure of potential adoption rate, or adoptability.

SECONDARY OUTCOMES:
To what extent are RA complication diagnoses actually affected by GenAI predictions? | Immediately after making the final diagnosis at discharge.
  Before patient discharge, physicians make final diagnoses and record which diagnosed complications or co-existing diseases were influenced by GenAI prediction information for each patient. The percentage of cases in which GenAI predictions affected the final diagnosis is calculated as a measure of AI's actual impact on routine diagnostic practice.

CONTACTS AND LOCATIONS:
Locations (1):
- Guang'anmen Hospital of China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Our previous study benchmarking LLMs for predicting a range of diseases. — https://pubmed.ncbi.nlm.nih.gov/38109889/
- See also: A recent paper reviewing LLMs in clinical decision support for autoimmune diseases. — https://www.nature.com/articles/s41584-025-01310-0